CLINICAL TRIAL: NCT01969396
Title: Evaluation of the Goldstein SonoBiopsy™ Catheter for Diagnosing Endometrial Pathology
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment considerations and current status of the clinical study
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 12-012
Record Dates: First submitted 2013-10-17; First posted 2013-10-25 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Menorrhagia; Endometrial Neoplasms; Polycystic Ovary Syndrome; Uterine Neoplasms
Keywords: Biopsy; Endometrial biopsy; Endometrial sampling; sonohysterography
MeSH Terms: conditions — Menorrhagia; Endometrial Neoplasms; Polycystic Ovary Syndrome; Uterine Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- SonoBiopsy Catheter (Experimental)
  Interventions: Device: SonoBiopsy Catheter
- Endometrial biopsy catheter (Active Comparator)
  Interventions: Device: Endometrial biopsy catheter

INTERVENTIONS:
Device: SonoBiopsy Catheter — Catheter utilized in dual role: sonohysterography and endometrial biopsy
  Other Names: Endometrial biopsy with sonohysterography
  Arms: SonoBiopsy Catheter
Device: Endometrial biopsy catheter — Endometrial sample obtained without the assistance of sonohysterography
  Other Names: Endometrial biopsy
  Arms: Endometrial biopsy catheter

SUMMARY:
To assess the adequacy of an endometrial biopsy sample obtained using sonohysterography.

ELIGIBILITY:
Inclusion Criteria:

* Patient with thickened endometrium
* Abnormal uterine bleeding

Exclusion Criteria:

* Pregnant
* Active pelvic infection
* Pelvic inflammatory disease
* Blood clotting disorders
* Sexually transmitted disease
* Uterine perforation
* Recent cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
percentage of adequate endometrial biopsies utilizing sonohysterography | 7 days
percentage of adequate endometrial biopsies collected without sonohysterography | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Mastellari, MD, Principal Investigator — Hospital Punta Pacifica
Locations (1):
- Hospital Punta Pacifica, Panama City, Panama